CLINICAL TRIAL: NCT00629031
Title: An Open Lable Randomised Two -Arm Study to Assess the Safety and Efficacy of Paromomycin Administered Intramuscularly at Two Different Dosing Regimens (14 Days Versus 21 Days) for the Treatment of Indian Visceral Leishmaniasis (VL)
Brief Title: An Open Lable Randomised Study to Assess the Safety and Efficacy of Short Course Paromomycin in Visceral Leishmaniasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Responsible Party: Shyam Sundar, Banaras Hindu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAMRC PSD
Record Dates: First submitted 2008-02-20; First posted 2008-03-05 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral leishmaniasis; Paromomycin
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Paromomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Paromomycin for 21 days @ 11mg/kg
  Interventions: Drug: Paromomycin
- 1 (Experimental): Paromomycin for 14 days @ 11mg/kg
  Interventions: Drug: Paromomycin

INTERVENTIONS:
Drug: Paromomycin — 11 mg/kg for 14 days
  Arms: 1
Drug: Paromomycin — Paromomycin for 21 days @ 11mg/kg by intramuscular injections

SUMMARY:
It is a randomized, double-blind, multi-center, two-arm study intended to assess the safety and efficacy of three different doses/dose regimens of paromomycin administered intramuscularly as follows: 11 mg/kg/day for 14 days and 11 mg/kg/day for 21 days for the treatment of visceral leishmaniasis (VL) in India.

DETAILED DESCRIPTION:
Paromomycin administered at a dose of 11 mg/kg/day IM for 21 days was previously demonstrated by iOWH and WHO to be as effective as amphotericin B administered IV at a dose of 1 mg/kg/every other day for a total for a total of 15 doses over 30 days in the treatment of VL in Bihar, India (protocol VLPM01) in a recently completed study (94.6% vs. 98.8% of subjects were disease free at 6 months, respectively). This new study is being conducted to determine whether similar or better efficacy and safety of IM paromomycin can be achieved with a shorter duration of treatment (14 days rather than 21 days) administered for a shorter duration (14 days rather than 21 days) than the regimen studied in the previous trial.

This shorter duration study will compare the initial and final cure (response to treatment) rates in subjects with VL receiving paromomycin at the following doses and dose regimens:

* Group A: paromomycin 11 mg/kg/day IM for 14 days
* Group B: paromomycin 11 mg/kg/day IM for 21 days

Because compliance generally improves with shorter duration of therapy, and better treatment compliance decreases the probability of the emergence of drug-resistant disease, administration of higher daily doses of paromomycin for a shorter time may improve efficacy without producing unacceptable toxicity. In addition, a treatment regimen of shorter duration would cost less and be easier to administer.

The current study is designed to explore different doses and dose regimens of IM paromomycin to determine the dose and dose regimen that should be recommended for first-line therapy for treatment of VL, while maintaining the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults, male or female, aged 5 to 55 years, inclusive, who have provided written informed consent.
* New or relapsed VL or prior VL treatment failure on a regimen not containing Paromomycin or AmBisome®. The diagnosis of VL must be confirmed by a parasite-positive splenic aspirate.

Exclusion Criteria:

* LFT greater than 3 times ULN ( AST, ALT, S.Bilirubin, Alkaline Phosphatase, Hb < 4 gm/dl.
* Platelet <40,000/ mm3
* Prothrombin Time > 3 Sec. longer than Control.
* Creatinine > 3 times

  * Normal Value For Male ( 0.6 to 1.1)
  * Normal Value For Female ( 0.5 to 0.9)
* Absolute Leucocyte count- < 1,000
* HIV infection
* Abnormal audiometric and/or vestibular dysfunction
* History of renal dysfunction
* Other severe medical conditions
* History of allergy or hypersensitivity to aminoglycosides
* Treatment with a parenteral aminoglycoside within 28 days prior to randomisation
* Previous VL treatment within the past 14 days
* Previous treatment for VL with paromomycin at any time
* Pregnancy, lactation, or lack of use of contraception in women of childbearing potential

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 329 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Final Cure | 6 months after the end of treatment

SECONDARY OUTCOMES:
Initial cure | End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Sundar, MD, Study Director — Banaras Hindu University
Locations (1):
- Kala-azar Medical Research Center, Rambag Road, Varanasi, India

REFERENCES:
- [Derived] Sundar S, Agrawal N, Arora R, Agarwal D, Rai M, Chakravarty J. Short-course paromomycin treatment of visceral leishmaniasis in India: 14-day vs 21-day treatment. Clin Infect Dis. 2009 Sep 15;49(6):914-8. doi: 10.1086/605438. PMID 19663597